CLINICAL TRIAL: NCT05118529
Title: Comparison of Physiological Response and Experience Between Sitting in Bed and Sitting in a Chair in Patients in Intensive Care
Brief Title: Physiological Response and Experience Between Sitting in Bed and Sitting in a Chair in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoU i VGR:275466
Record Dates: First submitted 2021-10-18; First posted 2021-11-12 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Intensive Care (ICU); Mobilization
Keywords: Immobilization; Intensive Care
MeSH Terms: interventions — Beds

STUDY DESIGN:
Intervention Model Description: Routine care vs additional mobilization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting in bed (Active Comparator): Sitting in bed with 60 degrees elevated back-rest during 20 minutes
  Interventions: Other: Routine care
- Sitting in chair (Experimental): Sitting in chair during 20 minutes
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Routine care — Mobilization to chair
  Other Names: Mobilization in bed

SUMMARY:
Background: In the work with early mobilization (EM), in intensive care, several types of EM are used A sitting in bed in semi- Fowler's position, sitting on the edge of the bed, and sitting in a chair. Nowadays, it is often possible to achieve a comfortable sitting in the beds in ICU. However, in a recent study by the same author group one of the findings was the importance to get out of bed. Getting out of bed was associated with decreasing feelings of hopelessness and being less ill. It also encouraged the will to fight for recovery.

There are few studies in intensive care that have examined what happens to circulation and oxygenation in various forms of sitting. Studies that examined the patient's own experience of sitting in bed compared to sitting in a chair are missing.

The aim is therefore to investigate physiological response and experience in patients in intensive care when sitting in bed or in a chair Method: Repeated measures randomized cross-over study Selection: Patients with respiratory and / or circulatory insufficiency requiring intensive care, Inclusion criteria: Approximately 30 respiratory and circulatory stable patients with emergency admission to intensive care. Aged over 18 years, who understands Swedish. The patient and / or relative are asked after the physician in charge has given medical approval. Recruitment is planned to be done by nurses in charge at the unit.

Exclusion criteria: Patients who have undergone planned surgery without complications.

Intervention: The participants in the study will be measured in two different positions; sitting in bed and sitting in chair. They are randomized to start either sitting in bed or in a chair and will sit for 20 minutes in each position, at 4 - hour intervals.

Data collection, physiological variables: The following physiological variables will be measured: Blood pressure and oxygenation by arterial needle and pulse by ECG. They will be measured before the intervention, at the beginning of the intervention, after ten minutes, at the end of the intervention and ten minutes afterwards Data collection, qualitative variables: Rating of the experience of exertion, pain and satisfaction.

Data analysis: Statistical analysis of differences between the two positions. For quantitative variables that are normally distributed, paired t-tests will be used. For qualitative variables and non-normally distributed quantitative variables, Wilcoxon character rank test or Mc Nemar test will be used

ELIGIBILITY:
Inclusion Criteria:

* emergency admission to intensive care
* age >18 years
* understanding Swedish

Exclusion Criteria:

* Respiratory or circulatory instability where mobilization is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
PaO2 | Within 8 hours after inclusion
  Arterial oxygen pressure
PaCO2 | Within 8 hours after inclusion
  Arterial carbon dioxide pressure

SECONDARY OUTCOMES:
Blood pressure | Within 8 hours after inclusion
  Systolic and diastolic pressure
SpO2 | Within 8 hours after inclusion
  Oxygen saturation
Perceived pain | Within 8 hours after inclusion.
  Visual analogue scale from 0-100 mm
Perceived exertion | Within 8 hours after inclusion
  Borg RPE scale from 6 to 20
Perceived satisfaction | Within 8 hours after inclusion
  Scale with 11 levels from 0 (no enjoyment) to 10 (maximum enjoyment).
Staff ratings of pain during mobilization | Within 8 hours after inclusion
  Visual analogue scale from 0-100 mm
Staff ratings of exertion during mobilization | Within 8 hours after inclusion
  Borg RPE scale from 6 to 20

CONTACTS AND LOCATIONS:
Locations (1):
- Göteborg University, Gothenburg, Sweden